CLINICAL TRIAL: NCT06360783
Title: Evaluation of a COVID-19 Quick Start "Test and Treat" Model in Africa
Brief Title: COVID-19 Quick Start - Test and Treat in Africa
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Duke Clinical Research Institute (Other); Clinton Health Access Initiative, Nigeria (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00111388
Record Dates: First submitted 2024-04-09; First posted 2024-04-11 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (5):
- Ghana: Aggregated testing and treatment data from centers in Ghana.
- Malawi: Aggregated testing and treatment data from centers in Malawi.
- Rwanda: Aggregated testing and treatment data from centers in Rwanda.
- Zambia: Aggregated testing and treatment data from centers in Zambia.
- Zimbabwe: Aggregated testing and treatment data from centers in Zimbabwe.

SUMMARY:
Duke University and the Clinton Health Access Initiative (CHAI), in partnership with the Ministries of Health (MoH) of Ghana, Malawi, Rwanda, Zambia, and Zimbabwe, aim to assess the implementation and impact of COVID-19 test -and -treat (T&T) demonstration programs

DETAILED DESCRIPTION:
Duke University and the Clinton Health Access Initiative (CHAI), in partnership with the Ministries of Health (MoH) of Ghana, Malawi, Rwanda, Zambia, and Zimbabwe, aim to assess the implementation and impact of COVID-19 test -and -treat (T&T) demonstration programs, titled "COVID-19 Quick Start Program". The MoHs in collaboration with CHAI will implement SARS-CoV-2 antigen testing programs linked to patient triage and initiation of eligible patients on a complete course of oral antivirals for COVID-19. The eligibility criteria and treatment regimens/duration may vary by country and over time depending on changes to guidelines.

This mixed method study will leverage data from three independent data collection activities to guide implementation:

1. Programmatic monitoring: A formative evaluation of the implementation of test and treat (T&T) programs to identify implementation gaps and help implementers make evidence-based decisions and course-correct as needed.
2. Collection of retrospective, patient-level data from treatment facility registers to understand impact of T&T implementation on testing and treatment initiation rates, as well as costs of treatment initiation for cost modeling.
3. Qualitative Semi-structured interviews with key stakeholders including MoH and public sector personnel, healthcare workers, and patients to understand the feasibility and acceptability of the program.

Data from this operational research study will help to ensure optimized delivery of T&T programs in low- and middle-income countries as the availability of therapeutics for COVID-19 scales up globally.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Able to provide informed consent
* Patients who have received COVID-19 testing and/or treatment at the facility
* Have a positive COVID-19 test and were prescribed oral antiviral medication (and may or may not have initiated on treatment (Only for subset of patients who will be followed to assess treatment completion and outcomes)

Exclusion Criteria:

None if other inclusion criteria are met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in participating countries who receive COVID testing and treatment at a participating facility.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Stakeholder Perspectives | up to 3 years
  Assess perspectives from key stakeholders including MoH and public sector personnel, healthcare workers, and patients on feasibility and acceptability of COVID-19 T&T programs as implemented

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Udayakumar, MD, Principal Investigator — Duke University
Locations (1):
- Duke Global Health Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Narayanasamy S, Gambanga F, Boeke CE, Udayakumar K, Brothers L, Wolfe CR, Agwuocha C, Asamoa-Amoakohene MN, Detleuxay K, Griffith BC, Hamza N, Joseph J, Kimani P, Kirungi R, Lufesi N, Mbewe N, McCarthy E, Mulenga M, Mukiibi M, Mwenifumbo T, Ofori-Boadu L, Okoli IU, Phongphila S, Regan S, Rwagasore E, Staple A, Tebor J, Tomno W, Umuraza S, Bosworth HB; COVID Treatment QuickStart Consortium Members; COVID-19 QuickStart Consortium Members. Mixed methods implementation research of oral antiviral treatment for COVID-19 in low- and middle-income countries: a study protocol. BMJ Open. 2025 Sep 18;15(9):e088465. doi: 10.1136/bmjopen-2024-088465. PMID 40973372